CLINICAL TRIAL: NCT02523807
Title: Tremor Monitoring Device
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Ilana Schlesinger, Director, Movement Disorders Institute, Rambam Health Care Campus
Other Study IDs: 0486-14-RMB
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Parkinson's Disease: Patients with tremor due to Parkinson Disease
- Patients with Essential tremor: Patients with tremor due to Essential tremor

SUMMARY:
Patients with tremor may have varying degrees of tremor at different times. The amplitude and frequency of tremor may change. The investigators observational study is intended to document this tremor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tremor due to Parkinson's disease or Essential tremor

Exclusion Criteria:

* Severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tremor due to Parkinson's disease or Essential tremor will be included
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum linear acceleration of the forearm. | Linear acceleration of the forearm will be measured for 15-60 minutes.
  We will measure linear acceleration of the forearm in meter per second squared.

SECONDARY OUTCOMES:
Maximum angular velocity of the forearm. | Maximum angular velocity of the forearm will be measured for 15-60 minutes.
  We will measure angular velocityof the forearm in degrees per second.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, M.D., Principal Investigator — Rambam Health Care Campus